CLINICAL TRIAL: NCT04593927
Title: Long Term Special Drug Use-results Surveillance for Mayzent in SPMS Patients (Prevention of Relapses and Delay of Progression of Physical Disability in Secondary Progressive Multiple Sclerosis)
Brief Title: Long Term Special Drug Use-results Surveillance for Mayzent in SPMS Patients
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CBAF312A1401
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Secondary Progressive Multiple Sclerosis (SPMS)
Keywords: Secondary Progressive Multiple Sclerosis; SPMS; Mayzent; Siponimod; Japan
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — siponimod

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mayzent: Patients administered Mayzent by prescription
  Interventions: Drug: Mayzent

INTERVENTIONS:
Drug: Mayzent — There is no treatment allocation. Patients administered Mayzent by prescription that have started before inclusion of the patient into the study will be enrolled.

SUMMARY:
This study is a single cohort, central registration system, all-case, open-label, multicenter observational study in patients using Mayzent for the indication of secondary progressive multiple sclerosis.

DETAILED DESCRIPTION:
This is a non-interventional study, and as such there is no binding treatment strategy, diagnosis/treatment procedures or visit schedule. The investigator should administer Mayzent as labelled. Routine medical practice will apply to visit frequency and evaluation variables, and only these data will be collected by the sponsor as part of the study procedures. The investigator should record data in the applicable CRFs at every visit if possible.

ELIGIBILITY:
Inclusion Criteria:

* Patients prescribed Mayzent for prevention of relapses and delay of progression of physical disability in secondary progressive multiple sclerosis

Exclusion Criteria:

-

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients using Mayzent for the following indication for a specified post-marketing period of time
  • Indication: prevention of relapses and delay of progression of physical disability in secondary progressive multiple sclerosis By allowing patients who started Mayzent administration before the conclusion of a contract for this study to be included in the study population after the contract, all patients treated with Mayzent will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 451 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AE), Serious Adverse Events (SAE) and Adverse Reactions | 24 months
  A SAE is defined as an AE whose description suggests that it is serious or whose outcome is fatal.
  An adverse reaction is defined as an adverse event that is suspected by the investigator to be causally related to Mayzent or whose causality is not recorded

SECONDARY OUTCOMES:
Physician's Global Assessment (PGA) of disease activity | month 12 and month 24
  Secondary Progressive Multiple Sclerosis (SPMS) symptom changes will be assessed an rated as "very much improved", "improved", "unchanged", "worsening" or "not assessable" in comparison with the symptoms at the start of Mayzent administration
Changes over time in Expanded Disability Status Scale (EDSS) score | Baseline, month 3, month 6, month 9, month 12, month 15, month 18, month 21 and month 24
  EDSS assesses disability. An overall score ranging from 0 (normal) to 10 (death due to MS) will be calculated.
Time to confirmed disability progression continuing for ≥ 3 months from the start of administration as assessed by the EDSS | 24 months
  Disability progression is defined as an increase of 1.5 points or more in patients with an EDSS score of 0 at baseline, an increase of 1 point or more in patients with an EDSS score of 0.5 to 5 at baseline and an increase of 0.5 points or more in patients with an EDSS score of 5.5 or more at baseline.
Time to confirmed disability progression continuing for ≥ 6 months from the start of administration as assessed by the EDSS | 24 months
  Disability progression is defined as an increase of 1.5 points or more in patients with an EDSS score of 0 at baseline, an increase of 1 point or more in patients with an EDSS score of 0.5 to 5 at baseline and an increase of 0.5 points or more in patients with an EDSS score of 5.5 or more at baseline.
Annual relapse rate | 24 months
  Annual relapse rate will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (143):
- Japan (143):
  - Novartis Investigative Site, Anjo, Aichi-ken
  - Novartis Investigative Site, Hekinan, Aichi-ken
  - Novartis Investigative Site, Ichinomiya, Aichi-ken
  - Novartis Investigative Site, Kariya, Aichi-ken
  - Novartis Investigative Site, Kasugai, Aichi-ken
  - Novartis Investigative Site, Nagakute, Aichi-ken
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Seto, Aichi-ken
  - Novartis Investigative Site, Hachinohe, Aomori
  - Novartis Investigative Site, Hirosaki, Aomori
  - Novartis Investigative Site, Ichihara, Chiba
  - Novartis Investigative Site, Ichikawa, Chiba
  - Novartis Investigative Site, Yachiyo, Chiba
  - Novartis Investigative Site, Tōon, Ehime
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Kurume, Fukuoka
  - Novartis Investigative Site, Gifu, Gifu
  - Novartis Investigative Site, Isesaki, Gunma
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Ōta, Gunma
  - Novartis Investigative Site, Fukuyama, Hiroshima
  - Novartis Investigative Site, Kure, Hiroshima
  - Novartis Investigative Site, Asahikawa, Hokkaido
  - Novartis Investigative Site, Hakodate, Hokkaido
  - Novartis Investigative Site, Iwamizawa, Hokkaido
  - Novartis Investigative Site, Kitami, Hokkaido
  - Novartis Investigative Site, Kushiro, Hokkaido
  - Novartis Investigative Site, Muroran, Hokkaido
  - Novartis Investigative Site, Rumoi, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Ako, Hyōgo
  - Novartis Investigative Site, Awaji, Hyōgo
  - Novartis Investigative Site, Itami, Hyōgo
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Nishinomiya, Hyōgo
  - Novartis Investigative Site, Hitachi, Ibaraki
  - Novartis Investigative Site, Hitachi-Naka, Ibaraki
  - Novartis Investigative Site, Toride, Ibaraki
  - Novartis Investigative Site, Tsuchiura, Ibaraki
  - Novartis Investigative Site, Tsukuba, Ibaraki
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Hanamaki, Iwate
  - Novartis Investigative Site, Ichinoseki, Iwate
  - Novartis Investigative Site, Kita-gun, Kagawa-ken
  - Novartis Investigative Site, Kagoshima, Kagoshima-ken
  - Novartis Investigative Site, Kamikoshikichō-oshima, Kagoshima-ken
  - Novartis Investigative Site, Ashigarakami, Kanagawa
  - Novartis Investigative Site, Atsugi, Kanagawa
  - Novartis Investigative Site, Hiratsuka, Kanagawa
  - Novartis Investigative Site, Isehara, Kanagawa
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Sagamihara, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Yokosuka, Kanagawa
  - Novartis Investigative Site, Nankoku, Kochi
  - Novartis Investigative Site, Kumamoto, Kumamoto
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Suzuka, Mie-ken
  - Novartis Investigative Site, Tsu, Mie-ken
  - Novartis Investigative Site, Kesennuma, Miyagi
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Miyakonojō, Miyazaki
  - Novartis Investigative Site, Chiisagata, Nagano
  - Novartis Investigative Site, Iida, Nagano
  - Novartis Investigative Site, Ina, Nagano
  - Novartis Investigative Site, Kitaazumi, Nagano
  - Novartis Investigative Site, Matsumoto, Nagano
  - Novartis Investigative Site, Nagano, Nagano
  - Novartis Investigative Site, Saku, Nagano
  - Novartis Investigative Site, Suwa, Nagano
  - Novartis Investigative Site, Sasebo, Nagasaki
  - Novartis Investigative Site, Kashihara, Nara
  - Novartis Investigative Site, Nagaoka, Niigata
  - Novartis Investigative Site, Niigata, Niigata
  - Novartis Investigative Site, Tsubame, Niigata
  - Novartis Investigative Site, Beppu, Oita Prefecture
  - Novartis Investigative Site, Ōita, Oita Prefecture
  - Novartis Investigative Site, Usa, Oita Prefecture
  - Novartis Investigative Site, Yufu, Oita Prefecture
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Ginowan, Okinawa
  - Novartis Investigative Site, Fujiidera, Osaka
  - Novartis Investigative Site, Higashiosaka, Osaka
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Ōsaka-sayama, Osaka
  - Novartis Investigative Site, Sakai, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Takatsuki, Osaka
  - Novartis Investigative Site, Saga, Saga-ken
  - Novartis Investigative Site, Ageo, Saitama
  - Novartis Investigative Site, Iruma-gun, Saitama
  - Novartis Investigative Site, Kawagoe, Saitama
  - Novartis Investigative Site, Koshigaya, Saitama
  - Novartis Investigative Site, Wako, Saitama
  - Novartis Investigative Site, Ohtsu-city, Shiga
  - Novartis Investigative Site, Ōmihachiman, Shiga
  - Novartis Investigative Site, Izumo, Shimane
  - Novartis Investigative Site, Fuji, Shizuoka
  - Novartis Investigative Site, Hamamatsu, Shizuoka
  - Novartis Investigative Site, Izunokuni, Shizuoka
  - Novartis Investigative Site, Oyama, Tochigi
  - Novartis Investigative Site, Shimotsuke, Tochigi
  - Novartis Investigative Site, Adachi City, Tokyo
  - Novartis Investigative Site, Adachi-ku, Tokyo
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Edogawa City, Tokyo
  - Novartis Investigative Site, Fuchū, Tokyo
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Itabashi Ku, Tokyo
  - Novartis Investigative Site, Kodaira, Tokyo
  - Novartis Investigative Site, Meguro City, Tokyo
  - Novartis Investigative Site, Nakano City, Tokyo
  - Novartis Investigative Site, Ōta-ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Kurayoshi, Tottori
  - Novartis Investigative Site, Toyama, Toyama
  - Novartis Investigative Site, Sakata, Yamagata
  - Novartis Investigative Site, Shimonoseki, Yamaguchi
  - Novartis Investigative Site, Shūnan, Yamaguchi
  - Novartis Investigative Site, Ube, Yamaguchi
  - Novartis Investigative Site, Akita
  - Novartis Investigative Site, Aomori
  - Novartis Investigative Site, Chiba
  - Novartis Investigative Site, Fukui
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Gifu
  - Novartis Investigative Site, Hiroshima
  - Novartis Investigative Site, Kagoshima
  - Novartis Investigative Site, Kochi
  - Novartis Investigative Site, Kumamoto
  - Novartis Investigative Site, Kyoto
  - Novartis Investigative Site, Nagasaki
  - Novartis Investigative Site, Niigata
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Ōita
  - Novartis Investigative Site, Saga
  - Novartis Investigative Site, Saitama
  - Novartis Investigative Site, Shizuoka
  - Novartis Investigative Site, Tokushima

IPD SHARING:
Plan to Share IPD: No